CLINICAL TRIAL: NCT02071940
Title: A Phase II Trial of PLX3397 in the Treatment of KIT Mutated Advanced Acral and Mucosal Melanoma
Brief Title: PLX3397 KIT in Acral aNd mucOsal Melanoma
Acronym: PIANO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Cancer Research UK (Other); Christie Charitable Funds (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11_DOG12_56
Record Dates: First submitted 2013-05-08; First posted 2014-02-26 (Estimated); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Malignant Melanoma
Keywords: Acral Melanoma subtypes; Mucosal Melanoma subtypes
MeSH Terms: conditions — Melanoma | interventions — pexidartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PLX3397 (Experimental): Patients will be given PLX3397 1000mg/day as monotherapy. Patients will remain on treatment as long as they are deriving benefit. This is a single cohort study and so there is no comparator arm - all patients receive the same treatment.
  Interventions: Drug: PLX3397

INTERVENTIONS:
Drug: PLX3397 — PLX3397 capsules 1000mg/day as monotherapy
  Other Names: Targeted therapy

SUMMARY:
KIT (receptor tyrosine kinase) mutations occur in 15% of acral and mucosal melanomas. PIANO is a single arm, phase II, open-label, multicentre study to evaluate the efficacy and safety (plus molecular basis of such effects) of the KIT inhibitor PLX3397 (developed by Plexxikon) in advanced KIT mutated acral and mucosal melanoma.

In this trial a total of 24 patients (9 in the first stage and 15 in the second stage) will receive treatment over a 24 month recruitment period.

Following consent and successful screening, patients will receive PLX3397 capsules 1000mg/day as monotherapy, and will remain on therapy as long as they are deriving clinical benefit. Patients will be seen every 4 weeks during treatment to monitor response and toxicity. Routine blood tests will be carried out at all visits and pharmacokinetics/pharmacodynamics sampling (1 x 8 milliliter(ml) whole blood sample) will be done pre-dose on Day 1 and Day 15, frozen and stored locally and sent to Plexxikon's vendor for central analysis at the end of the study. Imaging will be carried out every 12 weeks to monitor response. The first 9 patients will also receive two [18F]-fluorodeoxyglucose (FDG) PET scans (baseline and at Day 15).

From specific named participating sites, 12 patients will provide additional (optional) consent to take part in translational research. 5 of these patients will have a fresh tumour biopsy taken at baseline, at day 15 and upon disease progression. The same 5 patients plus an additional 7 patients (to give a total of 12 patients) will also donate blood samples at baseline, 2 weeks, 12 weeks and on disease progression for the evaluation of circulating tumour cells and circulating free tumour DNA.

All patients will be followed up every 6 months until death or for 12 months after the last patient has discontinued study treatment.

DETAILED DESCRIPTION:
The PIANO trial is an open-label, single-arm, multicentre phase II trial of PLX3397 in advanced acral and mucosal melanoma. All eligible patients will receive PLX3397 1000mg/day as monotherapy and will remain on treatment as long as they are deriving benefit (at the treating Investigator's discretion).

The primary objective of this study is to assess the efficacy of PLX3397 by review of the number of patients who are progression-free at 6 months. Additional objectives include assessing the safety of PLX3397, overall survival and (for a sub-set of patients) biomarker research.

A maximum of 24 eligible patients may be treated in this study. In order to recruit 24 patients, it is expected that a total of approximately 240 patients will need to be consented and screened for the KIT mutation, as only KIT mutant patients are eligible (and this is estimated to be 10-15% of this patient population). An interim analysis by the Independent Data Monitoring Committee will be done after 9 patients have been recruited and if less than 2 out of the 9 patients have demonstrated progression free survival at 6 months the trial will be terminated.

As only KIT mutant patients are eligible for inclusion, the very first step following consent is for patients' KIT mutation status to be tested. Only patients who have KIT mutations are eligible. Wherever possible, archival tissue samples taken at the time of diagnosis will be requested but if a suitable sample is not available or if following testing no result is obtained an additional fresh tumour sample would be collected via a biopsy. The tissue sample will be sent to specialist laboratories for KIT testing and the results of this test take 1-2 weeks. If the patient is found to have a KIT mutation which is not associated with PLX3397 resistance, they will return to clinic to complete the following study parameters and investigations upto 4 weeks prior to the start of treatment except those examinations which are marked with an (*) ;

* Demographic details
* Medical and surgical history including discussions of current medications
* Tumour evaluation according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria v1.1 using CT or MRI scans of the thorax, abdomen and pelvis within 28 days of scheduled start of treatment
* Vital signs and standard physical examination (to include blood pressure, pulse, temperature, height and weight)*
* Eastern Cooperative Oncology Group (ECOG) performance status*
* Laboratory investigations: full blood count, biochemistry (Urea & Electrolytes, creatinine, calcium, albumin, liver function tests, lactate dehydrogenase (LDH), glucose, phosphate) and clotting screen*
* Women of childbearing potential will have a urine or serum pregnancy test( within 72 hours of study entry)
* Electrocardiograph (ECG)*

If a patient undergoes a protocol-specified screening procedure as part of standard of care and the procedure occurs within 4 weeks then this data may be used for screening purposes and the test would not need to be repeated.

If the screening visit confirms that the patient is still eligible to take part in the study, they would return to clinic for a "baseline visit" and the following procedures would occur:

* Physical examination (including blood pressure and weight)
* Urine or serum pregnancy test in women of childbearing potential
* Electrocardiograph (ECG)
* ECOG Performance status
* Laboratory investigations: full blood count, biochemistry (U&Es, creatinine, calcium, albumin, liver function tests, LDH, glucose, phosphate) and clotting screen
* 1 x 8ml whole blood sample (Pharmacodynamics/pharmacokinetics (PK/PD)analysis) to be sent to Plexxikon's vendor for central analysis
* Adverse event (including treatment toxicity) assessments (see section 9.1 for definition of an adverse event).
* Review of concurrent medications
* PLX3397 prescription
* PET scan (first 9 patients only)

  * If the baseline visit is < 7 days since screening these investigations will not need to be repeated.

The patient would then return to clinic at day 15, day 29 (week 4), week 8 and then every 4 weeks in year 1 and every 8 weeks thereafter (until discontinuation of PLX3397). All visits have a window of +/- 3 days. The following procedures would be done at these visits:

* Physical examination (including blood pressure and weight).
* Electrocardiograph (ECG)
* ECOG Performance Status (PS)
* Laboratory investigations: full blood count, biochemistry (U&Es, creatinine, calcium, albumin, liver function tests, LDH, glucose, phosphate) and clotting screen.
* 1 x 8ml whole blood sample (PK/PD analysis) at Day 15 only (sent to Plexxikon's vendor for central analysis)
* Adverse event (including treatment toxicity) assessments until 30 days after discontinuation of PLX3397.
* Review of concurrent medications.
* Assessment of compliance with study medication.
* CT or MRI scans of the thorax, abdomen and pelvis at week 12, week 26 and every 12 weeks thereafter.
* Urine or serum pregnancy testing in women of childbearing potential on every visit ( except day 15 on treatment).
* PET scan after 2 weeks of therapy (day 15 ±3 days) - first 9 patients only

When the patient has discontinued the PLX3397 they then enter the follow-up phase of the study. Patients will be followed up until death or for 12 months after the last patient has discontinued study treatment. Patients can be followed up by telephone call every 6 months to assess current status and subsequent therapies. Alternatively follow-up can be in clinic especially in the case of complaints which may indicate late toxicity.

Translational Research

A subset of patients from named sites (The Christie National Health Service (NHS) Foundation Trust and The Royal Marsden NHS Foundation Trust) will also be asked to provide additional, optional consent to take part in translational research. 5 patients will have biopsies taken at 3 timepoints (baseline, at day 15 and on disease progression) and blood samples taken at 4 timepoints (baseline, at day 15, week 12 and on disease progression). In addition, a further 7 patients will give blood samples only (to give a total of 12 patients giving blood samples). Wherever possible translational blood samples will be taken at the same time as the standard trial blood samples which confirm that the patient is still eligible for study inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with KIT mutated histologically proven advanced mucosal or acral melanoma in which the mutation is not known to be associated with PLX3397 resistance
* Unresectable locally advanced or metastatic disease
* The presence of one or more clinically or radiologically measurable lesions at least 10mm in size
* ECOG performance status 0, 1 or 2
* Life expectancy greater than 12 weeks
* Age 18 or greater
* Women must be postmenopausal (no menstrual period for a minimum of 1 year) or have a negative serum pregnancy test on entry in the study (even if surgically sterilised). Men and women of childbearing potential must use adequate birth control measures for the duration of the study and should continue such precautions for 3 months after receiving the last dose of study treatment
* At least 28 days since major surgery and 7 days since skin/tumour biopsy
* Serum alanine transaminase (ALT) ≤2.5 x upper limit of normal (ULN) or serum aspartate aminotransferase≤2.5 x ULN
* Total serum bilirubin ≤1.5 x ULN
* Serum creatinine ≤1.5 x ULN
* Haemoglobin ≥90 g/L, absolute neutrophil count ≥1.5 x 109/L, platelets ≥100 x 109/L
* Prothrombin time (PT) ≤1.5 x ULN
* The ability to swallow and retain oral medication
* The capacity to understand the patient information sheet and the ability to provide written informed consent
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures

Exclusion Criteria:

* Intracranial disease, unless there has been radiological evidence of stable intracranial disease > 6 months. In the case of a solitary brain metastasis, evidence of a disease-free interval of at least 3 months post surgery. All patients previously treated for brain metastases must be stable off corticosteroid therapy for at least 28 days
* Women who are pregnant, nursing, or planning pregnancy within 6 months after the last treatment
* Men who plan to father a child within 3 months of the last treatment
* Use of any investigational drug within 30 days prior to screening
* Significant cardiac disease including patients who have or who are at significant risk of developing prolongation of corrected QT interval (QTc)
* Severe and/or uncontrolled medical disease
* Known chronic liver disease
* Known HIV infection
* Previous radiotherapy to 25% or more of the bone marrow and/or radiation therapy in the 4 weeks prior to study entry
* Prior exposure to a KIT inhibitor
* Patients with KIT mutations that are known to be associated with PLX3397 resistance
* Use of Chinese or herbal medication
* Any malabsorption syndrome (i.e. partial gastrectomy, small bowel resection, crohn's disease or ulcerative colitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-10; Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of PLX3397 | 6 months
  The primary objective of this study is to evaluate the efficacy of PLX3397 in KIT mutated advanced mucosal and acral melanoma as measured by the proportion of study participants tumour progression free at 6 months.

SECONDARY OUTCOMES:
Response rate | 12 weeks
  Patient's response rate is measured every 12 weeks (measured by CT scan) until confirmation of tumour progression or death and for a minimum period of 5 years in surviving patients.
Overall Survival | Participants are followed up for upto an average of 5 years or until the last patient dies, whichever comes first.
  Overall survival of patients is measured for a minimum of 5 years or until death, which ever comes first or 12 months after the last patient has progressed and finished treatment.
Safety of PLX3397 | minimum of 12 month following stoppage of treatment and for minimum of 5 years for patients remaining on treatment
  Safety of PLX3397 will be measured for a minimum of 12 months if patient discontinue treatment or diagnosed with disease progression and stop taking PLX3397 or for a minimum of 5 years in surviving patients receiving treatment. . Patients will be assessed for side effects at each clinic visit and all serious adverse events (SAEs)/ suspected unexpected serious adverse reaction (SUSARs) will be reported in accordance with applicable regulations.
Mechanism of response and resistance to PLX3397 | For 12 weeks or until the patient stops treatment
  Blood and tissue samples will be taken at specific timepoints in a subset of patients (additional consent required) to assess the mechanism of response and resistance to PLX3397. Patient samples are taken at baseline, week 2 and week 12 while on treatment or until patients are diagnosed with tumour progression at which point treatment stops.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Lorigan, MBBCH, FRCP, Principal Investigator — The Christie NHS Foundation Trust
Locations (8):
- United Kingdom (8):
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - The Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Abertawe Bro Morgannwg University Health Board, Singleton Hospital, Swansea, Wales
  - St James' University Hospital, Leeds, Yorkshire
  - Cancer Clinical Trials Centre- Weston Park Hospital, Sheffield, Yorkshire
  - Cambridge University Hospitals NHS FT - Addenbrookes Hospital, Cambridge
  - The Royal Marsden NHS Foundation Trust, London
  - Oxford University Hospitals NHS Trust- Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No
The output of the trial will be published in the peer review journals and scientific conferences